CLINICAL TRIAL: NCT02793388
Title: A Randomized Controlled Trial on Supervised Primaquine Use in Ethiopia
Brief Title: A Trial on Supervised Primaquine Use in Ethiopia
Acronym: SPRUE
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Menzies School of Health Research (Other)
Collaborators: Armauer Hansen Research Institute, Ethiopia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HREC 2016-2620
Record Dates: First submitted 2016-05-26; First posted 2016-06-08 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supervised primaquine arm (Active Comparator): Following standard schizontocidal treatment according to national guidelines and if haemoglobin levels are above 8g/dL and G6PD testing is normal, the patient receives primaquine (0.5mg/kg/day) for 14 days for radical cure. Supervision of primaquine is done on alternate days at home (attended by a home visitor) or at the health centre.
  Interventions: Drug: Supervised primaquine treatment
- Unsupervised primaquine arm (Active Comparator): Following standard schizontocidal treatment according to national guidelines and if haemoglobin levels are above 8g/dL and G6PD testing is normal, the patient receives primaquine (0.5mg/kg/day) for 14 days for radical cure for self administration.
  Interventions: Drug: Unsupervised primaquine treatment

INTERVENTIONS:
Drug: Supervised primaquine treatment — Following schizontocidal treatment malaria patients (P. falciparum and P. vivax) will receive 14days primaquine treatment if found to be G6PD normal. Primaquine treatment is provided supervised every other day.
  Arms: Supervised primaquine arm
Drug: Unsupervised primaquine treatment — Following schizontocidal treatment malaria patients (P. falciparum and P. vivax) will receive 14days primaquine treatment if found to be G6PD normal. Primaquine treatment is provided unsupervised.
  Arms: Unsupervised primaquine arm

SUMMARY:
This is a randomized, controlled, open label trial to assess the effectiveness of unsupervised versus supervised primaquine treatment in patients with uncomplicated malaria. In co-endemic regions, the risk of P. vivax relapse following treatment for P. falciparum is high. Hence patients infected with either P. vivax or P. falciparum will be included in the study. The study will be conducted in Ethiopia. Participants will be enrolled at health centres and provided with the recommended schizontocidal treatment plus primaquine radical cure which will be either supervised or unsupervised according to randomisation. Participants will be followed up for four months and assessed at regular intervals for the presence of patent and sub-patent malaria. The outcome of the study will contribute to an improved treatment scheme for uncomplicated malaria in this area.

ELIGIBILITY:
Inclusion Criteria:

* Fever (axillary temperature ≥37.5⁰C) or history of fever in preceding 48 hours
* Age >5 years
* Weight >5kg
* Written informed consent
* Living in the study area and willing to be followed for 4 months

Exclusion Criteria:

* General danger signs or symptoms of severe malaria (Appendix 17.1 and 17.2)
* Anaemia, defined as Hb <8g/dl
* Pregnant women as determined by Urine β-HCG pregnancy test
* Breast feeding women
* Known hypersensitivity to any of the drugs given
* Living in the same household as an individual enrolled into the study in the last 14 days

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
The incidence risk of symptomatic P. vivax malaria over 4 months in patients enrolled with P. vivax or P. falciparum malaria. | 4 months

SECONDARY OUTCOMES:
The incidence risk of symptomatic P. vivax malaria over 4 months in patients enrolled with P. vivax malaria infection. | 4 months
The incidence risk of symptomatic P. vivax malaria over 4 months in patients enrolled with P. falciparum malaria infection. | 4 months
The incidence rate of symptomatic P. vivax malaria over 4 months in patients enrolled with malaria due to P. falciparum or P. vivax. | 4 months
The incidence rate of symptomatic P. vivax malaria over 4 months in patients enrolled with P. vivax malaria. | 4 months
The incidence rate of symptomatic P. vivax malaria over 4 months in patients enrolled with P. falciparum malaria. | 4 months
The incidence risk of patent or sub-microscopic P. vivax malaria over 4 months in patients enrolled with malaria (sub-group analysis for patients recruited with P. vivax infection and P. falciparum infection) | 4 months
The incidence risk of any patent or sub-microscopic parasitaemia due to P. vivax or P. falciparum over 4 months in patients | 4 months
The cost-effectiveness of supervised primaquine therapy in terms of cost per malaria episode averted | 1 year
Socio-economic factors for adherence to primaquine treatment | 1 year
  Factors are collected through a semi-standardized questionaire. Factors include indicators for economic status, as well as information on educational background.

OTHER OUTCOMES:
The proportion of patients vomiting their medication within 1 hour of administration. | 1 day
The proportion of patients vomiting any of their primaquine doses during the 14 day supervised course. | 1 day
The proportion of adverse events and serious adverse events over 4 months in all patients. | 1 year
The incidence risk of severe anaemia (Hb<7g/dl) and/or the risk for blood transfusion over 4 months. | 4 months
The incidence risk of an acute drop in Hb >5g/dl within 14 days of starting primaquine treatment. | 14 days